CLINICAL TRIAL: NCT05258864
Title: Pilot Randomised Controlled Trial of an Online Personalised Normative Feedback Intervention to Reduce Drinking Among People With Unhealthy Alcohol Consumption
Brief Title: Pilot Trial of an Online Personalised Normative Feedback Intervention to Reduce Drinking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: HR-21/22-28339
Record Dates: First submitted 2022-02-17; First posted 2022-02-28 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-03

CONDITIONS: Alcohol Consumption
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Check Your Drinking (CYD) (Experimental): The CYD is a brief online intervention designed to provide personalized normative feedback aimed at motivating reductions in drinking
  Interventions: Behavioral: Check Your Drinking (CYD)
- Control (No Intervention): No Intervention Control

INTERVENTIONS:
Behavioral: Check Your Drinking (CYD) — The CYD is a brief online intervention designed to provide personalized normative feedback aimed at motivating reductions in drinking
  Arms: Check Your Drinking (CYD)

SUMMARY:
Unhealthy alcohol consumption is common in the UK and causes tremendous harm to the individual, as well as harm to others. A significant gap in providing alcohol support is that most people with unhealthy alcohol consumption will never receive advice to cut down on their drinking. However, many are interested in self-directed interventions to help them evaluate their drinking and to motivate reductions in alcohol use. One such promising intervention uses online personalised normative feedback (PNF) which compares a person's drinking with others in the general population of the same age and sex. PNF interventions are thought to work because many people with unhealthy alcohol consumption overestimate how much others drink. Multiple trials have demonstrated that providing PNF to people with unhealthy consumption reduces their alcohol use . While several UK websites do provide feedback on assessment of risk (e.g., Down Your Drink introductory section, Alcohol Change UK), there appears to be no online intervention that provides PNF for unhealthy alcohol consumption.

The major objective of this pilot project is to conduct a two-arm, parallel group randomised controlled trial (RCT) in which 1,318 participants recruited from the Prolific website who have identified themselves as drinking 14 or more units per week are randomly assigned to one of two groups - a) those who are offered a PNF report, and b) those in a no intervention comparator group. Participants in the comparator group will not be provided any intervention materials but will instead be given a list of the different components of the PNF feedback and will be asked to think about how useful they would find each of them. Follow-up assessment will occur at 1 and 6 months post-randomisation. The project is described as a pilot because it is a preliminary evaluation of the PNF intervention in a UK context.

ELIGIBILITY:
Inclusion Criteria:

Typically consume 14+ standard UK alcohol units per week Willingness to complete a 6-month follow-up survey 18 years of age or older

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1300 (Actual)
Dates: Start 2022-02-27 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Number of drinks consumed during a typical week | 6 months
  Number of drinks consumed during a typical week

CONTACTS AND LOCATIONS:
Locations (1):
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Available upon reasonable request from the senior author after publication of the results from the study.